CLINICAL TRIAL: NCT01909739
Title: The Effects of Statin on Postoperative Renal Function in Valvular Heart Surgery: a Randomized, Placebo-controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2013-0334
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2015-12

CONDITIONS: Acute Kidney Injury
Keywords: AKI, atrovastatin, Valvular heart surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Statin group (Experimental)
  Interventions: Drug: atrovastatin
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: atrovastatin — Atrovastatin 80mg was administered orally on the evening before surgery. Before anesthesia induction, atrovastatin 40mg was administered orally. And atrovastatin 40mg were administered orally in the evening of postoperative days 0, 1, and 2.
  Arms: Statin group
Drug: Placebo — Placebo 80mg was administered orally on the evening before surgery. Before anesthesia induction, placebo 40mg was administered orally. And placebo 40mg were administered orally in the evening of postoperative days 0, 1, and 2.
  Arms: Placebo group

SUMMARY:
The aim of this study is to examine the association between preoperative statin treatment and the incidence of postoperative acute kidney injury(AKI) in patients undergoing valvular heart surgery.

ELIGIBILITY:
Inclusion Criteria:

- patients over the age of 20 scheduled for valvular heart surgery

Exclusion Criteria:

1. Current statin use
2. Left ventricular ejection fraction < 30%
3. Preexisting congestive heart failure
4. Severe coronary artery disease
5. Hemodynamically unstable arrhythmia
6. Cardiogenic shock during perioperative period
7. Ventricular assist device
8. Severe renal dysfunction (eGFR < 15 ml/min per 1.73 m2)
9. History of liver disease or elevated serum transaminases
10. History of rhabdomyolysis or elevated creatinine kinase

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08-21 (Actual); Study Completion 2015-08-21 (Actual)

PRIMARY OUTCOMES:
Comparison of postoperative renal function with or without statin in patients undergoing valvular heart surgery | renal function change from 24-hour after surgery to 120-hour after surery
  BUN/Cr cystatin C eGFR urine output incidence of acute kidney injury(based on the AKIN criteria)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Park JH, Shim JK, Song JW, Soh S, Kwak YL. Effect of atorvastatin on the incidence of acute kidney injury following valvular heart surgery: a randomized, placebo-controlled trial. Intensive Care Med. 2016 Sep;42(9):1398-407. doi: 10.1007/s00134-016-4358-8. Epub 2016 Apr 27. PMID 27120082